CLINICAL TRIAL: NCT05798455
Title: Evaluation of the Safety and Efficacy of Sodium Pentaborate Pentahydrate in Patients With Advanced Renal Cell Carcinoma: An Open-label Single-arm Phase 1b/2 Trial
Brief Title: Evaluation of the Safety and Efficacy of Sodium Pentaborate Pentahydrate in Patients With Advanced Renal Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Principal Investigator, Tabriz University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 70926
Record Dates: First submitted 2023-03-11; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Sodium pentaborate pentahydrate
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sodium pentaborate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Capsules containing sodium pentaborate pentahydrate 500, 1000 and 1500 mg
  Interventions: Drug: Sodium Pentaborate

INTERVENTIONS:
Drug: Sodium Pentaborate — Capsules containing sodium pentaborate pentahydrate 500, 1000 and 1500 mg
  Other Names: Sodium pentaborate pentahydrate

SUMMARY:
This study investigates the safety and efficacy of sodium pentaborate pentahydrate in patients with advanced renal cell carcinoma.

DETAILED DESCRIPTION:
There is an increasing trend in the burden of renal cell carcinoma (RCC) globally. Although different therapies like tyrosine kinase inhibitors, ablative therapy, surgery, and immunotherapy have been suggested for RCC, they are not cost-effective. The present study will be conducted as an open-label, phase Ib/II study consisting of a dose-escalation stage followed by a cohort expansion stage. The trial will be conducted in the medical centers affiliated to the Tabriz University of Medical Sciences. Patients 18 years or older presenting with histologically confirmed RCC with a clear-cell component, that progressed to the advanced or metastatic stage will be recruited. The dose-escalation stage will determine the schedule and maximum tolerated dose (MTD) and/or recommended Expansion Stage dose of sodium pentaborate pentahydrate. One oral sodium pentaborate pentahydrate capsule once daily will be considered for evaluation in 21-day treatment cycles: 500 mg, 1000 mg, and 1500 mg. Subjects will accrue in escalation cohorts of 3-6 subjects using a "3 plus 3" design and dosing will begin at the 500 mg dose level of sodium pentaborate pentahydrate. During this stage, the decision to open a new cohort will be made when all subjects have been followed for at least 21 days following the first dose of sodium pentaborate pentahydrate(defined as the dose-limiting toxicity (DLT) Evaluation Period). In the dose-expansion stage, we will further assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of NaB in RCC using the recommended dose and schedule as determined in the dose-escalation stage. The primary objectives for the dose-escalation stage and dose-expansion stage will be to determine the maximum tolerated dose (MTD) and/or recommended dose and schedule for the subsequent expansion stage and to evaluate the preliminary efficacy of the sodium pentaborate pentahydrate by estimating the objective response rate, respectively. The investigator will assess each subject continuously to evaluate for potential new or worsening adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Histological confirmation of RCC with clear cell histology, including participants who may also have sarcomatoid features.
* Advanced (not amenable to curative surgery or radiation) or metastatic disease (American Joint Committee on Cancer [AJCC] stage IV)
* No prior systemic therapy for RCC with the following exception: one prior adjuvant or neoadjuvant therapy for fully resectable RCC if such therapy did not contain an agent targeting vascular endothelial growth factor (VEGF) or VEGF receptors and if at least 6 months after The last dose of adjuvant or neoadjuvant treatment has occurred.
* Karnofsky status score (KPS) 70%
* Measurable disease according to RECIST v1.1 according to the researcher
* Participants with favorable, moderate, and poor risk categories will be eligible for the study.
* Participants had to be stratified according to the International Metastatic RCC Database Consortium (IMDC) criteria according to favorable versus moderate versus poor risk status.
* Adequate hematologic and organ function, based on meeting all laboratory criteria within 14 days prior to the first dose of study treatment
* Patients who are willing and able to provide informed consent/written consent for the trial.
* Sexually active fertile patients and their partners must agree to use highly effective methods of contraception that alone or in combination with consistent and correct use during the study and for 5 months after the last dose of study treatment result in a lower failure rate. from 1% per year. An additional method of contraception, such as a barrier method (such as a condom), is recommended.
* A negative pregnancy test (urine or serum beta-human chorionic gonadotropin [β-hCG]) in screening sexually active women of childbearing potential.

Exclusion Criteria:

* Women who are pregnant, lactating, or planning to become pregnant within 3 months after the last dose of study drug and men who plan to father a child while enrolled in this study or within 5 months after the last dose of study drug.
* Any active central nervous system (CNS) metastases. Participants with treated and stable CNS metastases for at least one month were eligible.
* Any tumor that invades the superior vena cava (SVC), other major blood vessels, or the gastrointestinal tract. Any evidence of intratracheal or intrabronchial tumor
* Prior systemic therapy with VEGF, MET, AXL, KIT, or RET targeted therapy (including, but not limited to, sunitinib, pazopanib, axitinib, tivozanib, sorafenib, lenvatinib, bevacizumab, and cabozantinib)
* Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody, or any other antibody or drug that specifically co-stimulates T cells or Targets checkpoint routes.
* History of autoimmune disease requiring systemic therapy (eg, using disease-modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years.
* Diagnosis of immunodeficiency or receipt of systemic steroid or any other form of immunosuppressive therapy within two weeks prior to the first dose of trial therapy.
* Administration of a live, attenuated vaccine within 30 days before the first dose of study treatment.
* The patient has an uncontrolled or significant intercurrent disease
* Hematuria, hematemesis, or hemoptysis of more than 0.5 teaspoons (2.5 mL) of clinically significant red blood, or other histories of significant bleeding (eg, pulmonary hemorrhage) in the 12 weeks before the first dose.
* Cavity lung lesions or known manifestations of endobronchial disease.
* The lesion invades a major blood vessel including, but not limited to, the inferior vena cava, pulmonary artery, or aorta.
* Known psychiatric or substance abuse disorders that interfere with compliance with trial requirements.
* History or current evidence of any condition, treatment, or laboratory abnormality that may confound the results of the trial, interfere with the patient's participation throughout the trial, or in the opinion of the treating investigator is not in the patient's best interest for participation.
* The participant is currently participating in a study of another investigational agent and has received study treatment or used an investigational device within 4 weeks prior to the first dose of treatment.
* Allergy or previous hypersensitivity to the components of the studied therapeutic formulation has been identified. Patients with a history of infusion-related reactions to prior therapy may be eligible with sponsor approval if the reaction is considered mild and manageable with appropriate supportive care (eg, use of prodrugs per standard of care).
* Individuals with evidence of active malignancy other than RCC (except for curable early-stage cancer such as resected skin cancers and/or completely resected prostate cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-22 (Estimated); Primary Completion 2025-05-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and/or recommended dose | Day 21
  Determination of maximum tolerated dose (MTD) and/or recommended dose using Response Evaluation Criteria in Solid Tumors version 1.1
Objective response rate | Day 21
  Objective response rate using Response Evaluation Criteria in Solid Tumors version 1.1

SECONDARY OUTCOMES:
Duration of response | Days 0, 1, and 21
  Duration of response using Response Evaluation Criteria in Solid Tumors version 1.1
Progression free survival | Days 0, 1, and 21
  Progression free survival using Response Evaluation Criteria in Solid Tumors version 1.1
Disease control rate | Days 0, 1, and 21
  Disease control rate using Response Evaluation Criteria in Solid Tumors version 1.1
Overall survival | Days 0, 1, and 21
  Overall survival using Response Evaluation Criteria in Solid Tumors version 1.1
Adverse events | Days 0, 1, and 21
  Registration of adverse events in questionnaires using Response Evaluation Criteria in Solid Tumors version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Saeid Safiri, PhD, Principal Investigator — Tabriz University of Medical Sciences
Locations (1):
- Imam Reza hospital and Clinic of Salamat, Tabriz, East Azarbayejan, Iran

IPD SHARING:
Plan to Share IPD: No